CLINICAL TRIAL: NCT05400187
Title: The Effectiveness on Healthy Eating and Weight Management by Body Composition Assessment and Smart-phone Based Counselling Among Middle-aged Hong Kong Chinese: A 6-month Randomized Controlled Trial
Brief Title: Body Composition Assessment and Smart-phone Based Counselling on Healthy Eating and Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, XIE Yao Jie Grace, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P0013890
Record Dates: First submitted 2022-05-18; First posted 2022-06-01 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Weight Management; Healthy Diet
Keywords: Body Composition Assessment; Smart-phone Based Counselling; Weight Management; Health Eating Behavior; Middle-aged Hong Kong Chinese

STUDY DESIGN:
Intervention Model Description: The intervention group will receive a convenient body composition measurement and 6-month smart-phone based individualized counselling. Through close collaborations with the experts in nutrition, we can effectively disseminate the knowledge of weight management and control and healthy diet to the middle-aged population.
  No specific intervention will be given to the control group except the common anthropometric and body composition measurement.
Who Masked: Investigator, Outcomes Assessor
Masking Description: During the randomization session, the generated random numbers will be placed in opaque and tamperproof envelopes and sealed. Another independent person (other than statistician) will open all envelopes for eligible participants and responsible for arranging participants to undertake their corresponding treatments. Participants, investigators, and statistician will be concealed about the random allocation until each participant has been registered and the assignments have been made. The research assistant who will perform the outcome measures and the statistician are blinded to treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Body composition assessment and smart-phone based counselling group (Experimental): In this study, we consider body composition measurement together with an immediate brief counselling after the measurement as part of the intervention. The body composition measurement will allow the participants to get familiar with their own anthropometric data and serve as cues to actions of healthy diet adoption and weight management and control. Based on the measured body fat and anthropometric data, a trained research assistant will give brief individualized dietary and weight management counselling to the participants.
  The Whatsapp-based counselling and communication will heighten the awareness through reinforcing the need and benefits of body composition and weight control, the importance of energy balance, as well as providing professional and tailor-made advice on healthy eating and weight management. Qualitative dietary counselling will be offered every two weeks through the Whatsapp.
  Interventions: Behavioral: Body composition assessment and smart-phone based counselling
- Control group (No Intervention): Participants in the control group will receive the simple body composition measurement only, without an immediate counselling after the measurement. Whey will be informed the values of anthropometric data and body composition parameters, no detailed interpretation of the values will be delivered to them. They will also not receive the professional consultant of the healthy diet and weight management from the diatetitian during the intervention period.

INTERVENTIONS:
Behavioral: Body composition assessment and smart-phone based counselling — As for the body composition assessment, body fat and muscle thickness, body fat percentage and distribution will be measured and a brief face-to-face counseling soon after the measurement will be implemented to the participants. Body assessment were measured by the InBody 270 (Biospace, Seoul, Korea) device, which provides a convenient way of accurate body fat measurement comparable with those obtained using air displacement plethysmography (ADP) (about 90% precision).
  As for the Whatsapp-based counselling and communication session, qualitative dietary counselling will be offered every two weeks through the Whatsapp. One session contains 15 minutes, including the topics like making a balanced diet (55 % glucose, 30 % lipids and 15 % proteins), diversifying food intake, dietary advices and recommendations in healthy eating behaviors (e.g., eat slowly, eat at a regular time, avoid to skip a meal, drink at least 1.5 L of water each day).
  Arms: Body composition assessment and smart-phone based counselling group

SUMMARY:
This study proposed an integrated multi-disciplinary approach including a professional and convenient body composition measurement and an immediate counselling after the measurement, followed by 6-month smart-phone based individualized counselling. We believe that this approach will promote healthy eating behaviors and weight management among middle-aged Chinese in Hong Kong.

DETAILED DESCRIPTION:
This is a two-arm, individual level, 6-month randomized controlled trial. The intervention group will receive convenient body composition measurement and 6-month smart-phone based individualized counselling. No specific intervention will be given to the control group except the common anthropometric and body composition measurement. A pretest-posttest evaluation and between-group comparison will be used to test whether the impact/success of the project has been achieved.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand Cantonese and read Chinese;
* Self-reported vegetable and fruit consumption is less than 5 servings per day (one serving means 125 mL (½ cup) fresh, frozen or canned fruits or vegetables; or 250 mL (1 cup) raw leafy veggies or salad; or 125 mL (½ cup) 100% juice; or 1 fruit;
* Reachable by smart-phone and familiar with the use of smart-phone;
* Would not move from the local area during the study period.

Exclusion Criteria:

* Self-reported history of cardiovascular and pulmonary diseases, neurological disorder, musculo-skeletal disorder, osteoarthritis, and eating disorder;
* Receiving medically prescribed diet or physical activity intervention;
* For women, currently pregnant;
* Have been taking any medications or long-term supplement such as herbs;
* Cannot provide written informed consent.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The difference of the weight management belief | From baseline to 6 months after randomization
  Four items from belief domain of Chinese weight management scales (WMS) was used to measure the participants' belief of self weight management . Each item is measured by 3- or 4-point Likert scale. The total score change from 4 to 15 with higher scores indicating better weight management belief.
The difference of the weight management knowledge | From baseline to 6 months after randomization
  The knowledge of weight management was measured by 13 items from the general nutrition knowledge questionnaire (GNKQ). Each item carries one point for a correct answer and the maximum score is 13. A higher score shows better weight management knowledge.

SECONDARY OUTCOMES:
The difference of health eating behavior | From baseline to 6 months after randomization
  Respondents' food knowledge and behavior were obtained through the food behavior questionnaire (FBQ). The FBQ is a questionnaire with 18 questions querying respondents' behaviors and knowledge about various areas of food and diet-related health such as nutrition label reading behaviors, knowledge of diet/disease relationships and some meal consumption patterns.
Weight | From baseline to 6 months after randomization
  Weight in kg.
Body mass index (BMI) | From baseline to 6 months after randomization
  BMI in kg/m^2
Waist circumference | From baseline to 6 months after randomization
  Waist in cm
Hip circumference | From baseline to 6 months after randomization
  Hip in cm
Thigh circumference | From baseline to 6 months after randomization
  Thigh in cm
Systolic blood pressure | From baseline to 6 months after randomization
  Systolic blood pressure in mmHg
Diastolic blood pressure | From baseline to 6 months after randomization
  Diastolic blood pressure in mmHg
Body fat percentage | From baseline to 6 months after randomization
  Body fat percentage was measured by a professional body composition analyzer named InBody 270 in %.
Body fat mass | From baseline to 6 months after randomization
  Body fat mass was measured by a professional body composition analyzer named InBody 270 in kg.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Jie Xie, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Hong Kong

REFERENCES:
- [Derived] Yang Q, Zhang Y, Liang J, Wang HH, Ma T, Qin J, Xie YJ. Nurse-led counselling and smartphone-based coaching for dietary behaviors, weight management and cardiometabolic risk in middle-aged Chinese in Hong Kong: a randomized controlled trial. Eur J Cardiovasc Nurs. 2026 Jan 29:zvag027. doi: 10.1093/eurjcn/zvag027. Online ahead of print. PMID 41605251